CLINICAL TRIAL: NCT04398056
Title: Chemotherapy Plus Subsequent Loco-regional Radiotherapy Combined With Toripalimab for the de Novo Metastatic Nasopharyngeal Carcinoma: a Single Center, Phase II Clinical Trial.
Brief Title: Chemotherapy Plus Subsequent Loco-regional Radiotherapy Combined With Toripalimab in the De Novo Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, professor & chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC2019
Record Dates: First submitted 2020-05-06; First posted 2020-05-21 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: de novo nasopharyngeal carcinoma; radiotherapy; PD-1
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Drug Therapy; Radiotherapy; toripalimab

STUDY DESIGN:
Intervention Model Description: This study used Simon's two-stage design. The main purpose of the study was to determine the objective response rates (PR+CR) of local-regional radiotherapy combined with Toripalimab followed by systemic chemotherapy for de novo metastatic nasopharyngeal carcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy plus radiotherapy and Toripalimab (Experimental): Patients were treated with PF chemotherapy for a maximum of six cycles followed by loco-regional radiotherapy combined with toripalimab.
  Interventions: Drug: Chemotherapy plus radiotherapy and Toripalimab

INTERVENTIONS:
Drug: Chemotherapy plus radiotherapy and Toripalimab — 1. Chemotherapy:
     The PF regimen included 5 g/m2 5-fluorouracil via a continuous intravenous infusion over 120 h and an intravenous administration of 100 mg/m2 cisplatin on day 1 for a maximum of six cycles.
  2. Radiotherapy, intensity-modulated radiation therapy (IMRT), PTVnx:66-70Gy/30-33F; PTVnd:66～70Gy/30～33F; PTV1:60～64Gy/30～33F; PTV2:50～54Gy/30～33F, 5 fractions per week, for 6 weeks
  3. Toripalimab 240mg every three weeks (Q3W) began on the first day of radiotherapy until an intolerable toxicity, or disease progression, or withdrawal of consent, or the investigator determines that he or she has to withdraw from treatment, or has been treated for up to 2 years.

SUMMARY:
The purpose of this study is to preliminarily evaluate the efficacy and safety of chemotherapy plus subsequent loco-regional radiotherapy combined with toripalimab for the de novo metastatic nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a single center , single arm, phase II study. All eligible patients with the de novo metastatic NPC are treated with chemotherapy plus subsequent loco-regional radiotherapy combined with toripalimab. The primary objective of this study is to assess objective response rate of chemotherapy plus subsequent loco-regional radiotherapy combined with toripalimab in de novo metastatic nasopharyngeal carcinoma . The secondary objective is to assess progression free survival, and Adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Had histopathologically confirmed metastatic NPC that was diagnosed as stage IVb NPC as defined by the AJCC, 8th edition;
2. Patients evaluated to have a complete response (CR) or partial response (PR) by an imaging study after three cycles of cisplatin plus 5-fluorouracil (PF) chemotherapy;
3. Patients who did not receive any previous systemic chemotherapy;
4. Patients with a Karnofsky performance status (KPS) score of at least 70;
5. Patients with adequate organ function (white blood cell count of at least 4.0x109 per L; absolute neutrophil of at least 2.0x109 per L; hemoglobin concentrations of at least 90 g/L; platelet cell count of at least 100 x109 per L; aspartate transaminase and alanine transaminase levels less than 2.5 times the upper limit of the normal value; and creatinine clearance rate of at least 60 mL/min);
6. Patients who provided written informed consent;
7. Patients who agree to regular follow-up visits.

Exclusion Criteria:

1. Patients with recurrent mNPC who received prior definitive radiotherapy/chemoradiotherapy;
2. Patients with life-threatening medical disorders;
3. Patients who were pregnant or breastfeeding;
4. Patients with other invasive malignant diseases within the past 5 years, other than excised basal-cell skin carcinoma, cervical carcinoma in situ, superficial bladder tumors (Ta, Tis, and T1);
5. Patients with serious comorbidities.
6. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Subjects with the following conditions will not be excluded from this study: asthma that requires intermittent use of bronchodilators, hypothyroidism stable on hormone replacement, vitiligo, Graves' disease, or Hashimoto's disease. Additional exceptions may be made with medical monitor approval;
7. Known history of hypersensitivity to any components of the Toripalimab formulation;
8. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed;
9. Active central nervous system (CNS) metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease);
10. Uncontrolled clinically significant medical condition, including but not limited to the following:

    1. congestive heart failure (New York Health Authority Class > 2);
    2. unstable angina;
    3. myocardial infarction within the past 12 months;
    4. clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
11. Active infection or an unexplained fever; 38.5℃ during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled);
12. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease;
13. Any other medical (eg, pulmonary, metabolic, congenital, endocrinal, or CNS disease), psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results;
14. Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation based on institutional guidelines and tests. Testing may include the following: HBV DNA, HCV RNA, hepatitis B surface antigen, or anti-Hepatitis B core antibody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1 year
  The proportion of patients who achieved an objective response, defined as those with radiologically confirmed complete or partial response according to RECIST 1.1 assessed by the investigator;

SECONDARY OUTCOMES:
Disease Control Rate | 1 year
  The proportion of patients who achieved disease control, defined as those with RECIST-defined objective response or stable disease
Progression-free survival | 1 year
  The time is defined from the enrolment to RECISTdefined progression or death from any cause
The toxicity grade will be assessed according to CTCAE 5.0. | 1 year
  Safety profiles

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen SY, Duan XT, Li HF, Peng L, Wang ZQ, Xu GQ, Hua YJ, Zou X, You R, Ouyang YF, Liu YP, Gu CM, Yang Q, Jiang R, Zhang MX, Lin M, Xie YL, Lin C, Ding X, Xie RQ, Duan CY, Zhang WJ, Huang PY, Chen MY. Efficacy of sequential chemoradiotherapy combined with toripalimab in de novo metastatic nasopharyngeal carcinoma: A phase II trial. Cell Rep Med. 2023 Nov 21;4(11):101279. doi: 10.1016/j.xcrm.2023.101279. Epub 2023 Nov 10. PMID 37951218